CLINICAL TRIAL: NCT06553495
Title: A Comparative Analysis of Intertransverse Nerve Block and Paravertebral Nerve Block in Endoscopic Hepatectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Chen (Other)
Responsible Party: Sponsor-Investigator, Jie Chen, 临床教授, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-098
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intertransverse nerve block (Experimental): To study the analgesic effect of intertransverse nerve block after endoscopic hepatectomy
  Interventions: Other: Nerve block
- paravertebral nerve block (Placebo Comparator): To study the analgesic effect of paravertebral nerve block after endoscopic hepatectomy
  Interventions: Other: Nerve block

INTERVENTIONS:
Other: Nerve block — Analgesic effect of different nerve blocks

SUMMARY:
This study aims to compare the analgesic effect of intertransverse nerve block and paravertebral nerve block after endoscopic hepatectomy, evaluate its effectiveness and safety, and provide new ideas and clinical basis for postoperative pain management of liver surgery.

DETAILED DESCRIPTION:
This study was a prospective, double-blind, randomized controlled trial. Patients who were eligible for laparoscopic partial liver resection in our center were included, with intertransverse nerve block as the experimental group and paravertebral nerve block as the control group. Through the analysis of postoperative pain score 30min to 24h, the number of effective analgesic pump compressions within 24h, the amount of analgesic drugs used, complications and other data, To evaluate the efficacy and safety of intertransverse nerve block in patients undergoing laparoscopic partial liver resection.

ELIGIBILITY:
Inclusion Criteria:1:

1.18-80 years old adult, BMI<27.9kg/m2

2: 2. American Society of Anesthesiologists ASA Grade I-III

3: 3. Patients with laparoscopic partial liver resection such as liver tumors

4: 4. Willing to participate in this study and sign the informed consent form

-

Exclusion Criteria:

1. 1. The patient or family member refuses to sign the informed consent form
2. 2. Blood coagulation dysfunction, local infection
3. 3. Those who have communication, communication disorders or mental abnormalities
4. 4. Patients with severe heart, pulmonary and renal insufficiency or patients with central system diseases
5. 5. For any reason, it cannot be matched with the study or the researcher believes that it is not appropriate to be included in this experiment.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of effective compressions of the analgesic pump within 24 hours after surgery | Within 24 hours after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No